CLINICAL TRIAL: NCT01505439
Title: A Prospective, Open Label, Single Arm, Multicenter Study to Estimate the Efficacy and Safety of Solifenacin in Female With Clinically Significant Stress Urinary Incontinence and Urgency Urinary Incontinence
Brief Title: A Study to Estimate the Efficacy and Safety of Solifenacin in Female With Stress Urinary Incontinence and Urgency Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeong Gu Lee (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jeong Gu Lee, Professor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VENUS-MUI
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Stress Urinary Incontinence; Urgency Urinary Incontinence
Keywords: solifenacin; bladder symptom
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solifenacin group (Experimental): Once daily
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: solifenacin — oral
  Other Names: Vesicare

SUMMARY:
This study is to investigate the effects of solifenacin on urgency urinary incontinence symptoms and incontinence quality-of-life (I-QoL) in female patients with clinically significant stress urinary incontinence accompanied by urgency urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patients are selected from those who meets one of criteria
* Patients with a positive cough provocation test
* Based on 3-day voiding diary, patients with:

  * Urinary frequency (eight or more micturitions per day or 24 hours)
  * Urinary urgency (two or more episodes per day or 24 hours)
  * Urge incontinence (three or more episodes for 3 days)

Exclusion Criteria:

* Breast-feeding women or females of childbearing potential with the intention to become pregnant during the study
* Post-void residual urine volume (PRV) of 150 cc or more
* Patients who experienced acute ureteral obstruction requiring an indwelling catheter
* Patients who experienced clinically significant pelvic organ prolapse or lower urinary tract surgery within 6 months prior to the initiation of the present study
* Patients who underwent a urinary incontinence operation within 1 year
* Any condition that, in the opinion of the investigator, is a contraindication for anticholinergic treatment, including severe narrow-angled glaucoma, urinary retention, gastric retention, severe myasthenia, severe hepatic insufficiency or severe ulcerative colitis
* Significant hepatic or renal disease, defined as having greater than twice the upper limit of the reference ranges for serum concentrations of aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase or creatinine
* Patients who have any of neurological disorders such as stroke, multiple sclerosis, spinal cord injury, and Parkinson's disease
* Patients who use an indwelling catheter or practice intermittent self-catheterization
* Recurrent UTIs defined as having been treated for symptomatic UTIs 3 times or more in the last year
* Symptomatic acute urinary tract infection (UTI) during the run-in period
* Patients who received any of the following prohibited concomitant drugs within 14 days prior to randomization: Treatment performed within the 14 days preceding randomization, or expected to initiate treatment during the study with:

  * Any anticholinergics other than the trial drug
  * Any drug treatment for overactive bladder. Estrogen treatment started more than 2 months prior to inclusion is allowed
* Patients taking an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
* Patients with chronic constipation or history of severe constipation
* Treatment with any of potent CYP3A4 inhibitors, such as cyclosporine, vinblastine, macrolide antibiotics (e.g. erythromycin, clarithromycin, azithromycin) or antifungal agents (e.g. ketoconazole, itraconazole, micronazole)
* Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to study initiation and not agreeing to use such methods during the entire study period and for at least 1 month thereafter. Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives, surgical procedures (tubal ligation or vasectomy), or continence
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in the number of urge urinary incontinence episodes per 24 hours between baseline and week 12 | Baseline and week 12

SECONDARY OUTCOMES:
Percent change in the mean number of urge urinary incontinence episodes per 24 hours | Baseline, week 4 and week 12
Change in the mean number of urge urinary incontinence episodes per 24 hours | Baseline, week 4 and week 12
  urgency episodes: defined as those with a Bladder Sensation Scale rating of ≥ 3 in the voiding diary
Change in the mean frequency of urination per 24 hours | Baseline, week 4 and week 12
Percent change in the mean frequency of urination | Baseline, week 4 and week 12
Changes in the mean and sum rating on the Bladder Sensation Scale per 24 hours | Baseline, week 4 and week 12
Change in the mean number of severe urgency episodes per 24 hours | Baseline, week 4 and week 12
  severe urgency episodes: defined as those with a Bladder Sensation Scale rating of ≥ 4 in the voiding diary
Changes in overactive bladder symptom score (OABSS) questionnaire | Baseline, week 4 and week 12
  Change in total and each of OABSS items
Changes in short urogenital distress inventory (UDI-6) | Baseline, week 4 and week 12
  Change in total and each UDI-6 items
Changes in short incontinence impact questionnaire (IIQ-7) | Baseline, week 4 and week 12
  Change in total and each of IIQ-7 items
Safety assessed by the incidence and severity of side effects | For 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Site KR00003, Daegu
  - SIte KR00004, Incheon
  - Site KR00001, Jeonam
  - Site KR00002, Jungnam
  - Site KR00005, Pusan
  - Site KR00006, Seoul